CLINICAL TRIAL: NCT04348045
Title: MAZEPPA: Phase II PRODIGE-GERCOR Study to Evaluate MAintenance Therapy With Olaparib or Selumetinib Plus Durvalumab According to BRCAness and KRAS Somatic Status Personalized in Metastatic Pancreatic Adenocarcinoma Patients
Brief Title: Maintenance With Olaparib or Selumetinib + Durvaluma for m-PDAC Guided by BRCAness and KRAS Status.
Acronym: MAZEPPA
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: GERCOR - Multidisciplinary Oncology Cooperative Group (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: MAZEPPA D19-02 PRODIGE-72
Record Dates: First submitted 2020-04-08; First posted 2020-04-15 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Metastatic Pancreatic Adenocarcinoma
Keywords: BRCAness status; KRAS somatic status
MeSH Terms: interventions — olaparib; AZD 6244; durvalumab; Leucovorin; Fluorouracil; Irinotecan

STUDY DESIGN:
Intervention Model Description: Patients with a BRCAness somatic profile: olaparib Arm A. Patients with no BRCAness profile and with KRAS mutation randomization between durvalumab plus selumetinib Arm B, versus FOLFIRI Arm C.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ARM A - olaparib (Experimental): Olaparib tablets at 300 mg orally twice daily until PD (RECIST 1.1) or unacceptable toxicity.
  Interventions: Drug: Arm A - Olaparib
- ARM B - durvalumab plus selumetinib (Experimental): Durvalumab plus selumetinib until PD (RECIST 1.1 and/or iRECIST), unacceptable toxicity, withdrawal of consent, or death.
  Durvalumab administered IV at a flat dose of 1500 mg on day 1 of every 28-day cycle,
  Selumetinib administered as 75 mg twice daily dose for 21 days on and 7 days off (a 28-day cycle).
  Interventions: Drug: ARM B - durvalumab plus selumetinib
- ARM C - FOLFIRI (Active Comparator): FOLFIRI FOLFIRI (irinotecan 180 mg/m2 IV on day 1, folinic acid 400 mg/m2 IV on day 1, 5-FU 400 mg/m2 IV bolus on day 1 and 2, and 46h IV infusion of 5-FU 2400 mg/m2 every 2 weeks) until PD (RECIST 1.1) unacceptable toxicity, withdrawal of consent, or death.
  Interventions: Drug: ARM C FOLFIRI

INTERVENTIONS:
Drug: Arm A - Olaparib — 300 mg orally twice daily, for a total daily dose of 600mg
  Study treatment can be dose-reduced to :
  First step : 250 mg twice daily , for a total daily dose of 500 mg Second step: 200 mg twice daily taken twice daily, for a total daily dose of 400 mg No further dose reduction is allowed, and study treatment should be discontinued.
  Other Names: AZD-2281
  Arms: ARM A - olaparib
Drug: ARM B - durvalumab plus selumetinib — Durvalumab administered IV at a flat dose of 1500 mg on day 1 of every 28-day cycle, Selumetinib Starting Dose : 75 mg twice daily
  Study treatment can be dose-reduced to :
  Dose Level -1 : 75 mg once daily Dose Level -2 : 50 mg twice daily Dose Level -3 : 50 mg once daily
  Other Names: MEDI-4736 plus AZD-6244
  Arms: ARM B - durvalumab plus selumetinib
Drug: ARM C FOLFIRI — FOLFIRI every two weeks Irinotecan 180 mg/m2 Intravenous (IV) on day 1 Folinic acid 400 mg/m2 IV on day 1, 5-FU 400 mg/m2 IV bolus on day 1 and 2, and 46h IV infusion of 5-FU 2400 mg/m2
  Other Names: folinic acid, fluorouracil, and irinotecan
  Arms: ARM C - FOLFIRI

SUMMARY:
MAZEPPA is open-label, phase II study to assess the efficacy of a genomic-driven maintenance therapy in terms of PFS in Pancreatic ductal adenocarcinoma (PDAC) patients with disease controlled after 4 months of mFOLFIRINOX chemotherapy as following:

Patients with a BRCAness somatic profile: olaparib Arm A. Patients with no BRCAness profile and with KRAS mutation randomization between durvalumab plus selumetinib Arm B, versus FOLFIRI Arm C.

DETAILED DESCRIPTION:
Searching for efficient maintenance therapies in metastatic PDAC patients whose disease has been controlled using an induction chemotherapy is crucial for two main reasons:

1. Patients may stop IV toxic chemotherapy while their tumor remains under control. Although up to 70% of PDAC patients achieve tumor control when treated during induction with mFOLFIRINOX, toxicity of this regimen, particularly neuropathy and fatigue, remains a key concern.
2. Tumor control may be extended, which might improve quality of life (QoL) and survival.

Patients are included in MAZEPPA study based on the genetic profile of their tumor.

* If a BRCA gene mutation is present in the tumor, treatment with the drug olaparib will be proposed (arm A), regardless of the status of the other genes analyzed.
* In the absence of a mutation in the BRCA gene and in the presence of a mutation in the KRAS gene, a treatment combining immunotherapy and targeted therapy (durvalumab and selumetinib - Arm B) or chemotherapy by FOLFIRI (arm C) will be proposed.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated informed consent,
2. Age ≥18 years
3. Body weight >30 kg,
4. Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up,
5. Life expectancy of at least 4 months,
6. Eastern Cooperative Oncology Group Performance Status (ECOG PS) 0-1,
7. Pathologically confirmed pancreatic adenocarcinoma with distant metastases (stage IV disease),
8. No prior therapy for metastatic disease other than mFOLFIRINOX (in case of previous adjuvant therapy, the interval between the end of adjuvant chemotherapy and relapse must be >6 months),
9. Stability or tumor response (Response evaluation criteria in solid tumors [RECIST] 1.1) after 4 months of mFOLFIRINOX (8 cycles) for metastatic disease,
10. Have tissue from archival tissue sample from surgery or biopsy identified and confirmed as available for study
11. Availability of tumor somatic genetic analyses data, performed during the first 4 months of mFOLFIRINOX (specific informed consent),
12. In case of germinal BRCA gene mutation identified before inclusion the patient can be included until olaparib receives a marketing authorization for the treatment indication of the patients in the study and the treatment is available in the retail pharmacy; it will be prescribed according to the summary product characteristics (SmPC),
13. At least one measurable or evaluable lesion as assessed by CT-scan or MRI according to RECIST 1.1 and feasibility of repeated radiological assessments,
14. Normal organ and bone marrow function prior to administration of study treatment as defined below:

    * Hemoglobin ≥ 10.0 g/dL with no blood transfusion in the past 28 days,
    * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L,
    * Platelet count ≥ 100 x 109/L,
    * Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN),
    * Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) ≤ 2.5 x institutional ULN unless liver metastases are present in which case

      ≤ 5x ULN,
    * Creatinine clearance (CrCl) ≥ 50 mL/min estimated using the Cockcroft-Gault equation, Estimated CrCl =(140-age [years]) x weight (kg) (x F)a serum creatinine (mg/dL) x 72 a F=0.85 for females and F=1 for males.
15. Absence of known dihydropyrimidine dehydrogenase (DPD) deficiency,
16. Female patients must be surgically sterile, or be post-menopausal, or have negative serum pregnancy test if pre-menopausal at inclusion and must commit to using reliable and appropriate methods of contraception during the study and during at least 6 months after the end of studytreatment (when applicable).

    Women will be considered post-menopausal if they have been amenorrhoeic for 12 months without an alternative medical cause. The following age-specific requirements apply:
    * Women < 50 years of age would be considered post-menopausal if they have been amenorrhoeic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone (LH) and follicle-stimulating hormone (FSH) levels in the postmenopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy).
    * Women ≥ 50 years of age would be considered post-menopausal if they have been amenorrhoeic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses > 1 year ago, had chemotherapy-induced menopause with last menses > 1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy). All female patients with reproductive potential must have a negative pregnancy test (beta human chorionic gonadotropin [β-HCG]) within 72 hours prior to starting the protocol treatment. Breastfeeding is not allowed. Male patients must agree to use effective contraception in addition to having their partner use a contraceptive method as well during the trial and during at least 6 months after the end of the study treatment. Men and women with childhood potential are required to use adequate birth control during the study,
17. Registration in a national health care system (PUMa; Couverture Maladie Universelle included).

Exclusion Criteria:

1. Histology other than PDAC
2. Toxicities after mFOLFIRINOX treatment not resolved to ≥ grade 1 prior to maintenance treatment, except for oxaliplatin induced neuropathy, alopecia, or grade ≥ 2 are permitted
3. Patients with known brain metastases at inclusion,
4. Enrollment in another therapeutic trial
5. Evidence of interstitial lung disease, any active non-infectious pneumonitis, or known active infection including active tuberculosis
6. Hepatitis B virus (HBV; known positive HBV surface antigen (HbsAg) result), hepatitis C virus (HCV), or human immunodeficiency virus (positive HIV ½ antibodies).
7. Active uncontrolled infection, current unstable, or uncompensated respiratory or cardiac conditions, or active digestive hemorrhages less than 3 months,
8. Patient has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the study,
9. Live vaccine administration within 30 days prior to the first dose of study treatment,
10. Treatment with any other investigational medicinal product within 28 days prior to study entry,
11. Other malignancy unless curatively treated with no evidence of disease for ≥ 5 years except: adequately treated non-melanoma skin cancer, curatively treated in situ cancer of the cervix, ductal carcinoma in situ (DCIS), and stage 1, grade 1 endometrial carcinoma,
12. Uncontrolled intercurrent illness, including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, acute coronary syndrome within 6 months prior to starting treatment, prior or current cardiomyopathy, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent,
13. Resting electrocardiogram (ECG) indicating uncontrolled, potentially reversible cardiac conditions, as judged by the Investigator or patients with congenital long QT syndrome. Mean corrected QT interval (QTc) for heart rate using the QTcF formula ≥ must be <470 ms,
14. Pregnancy/lactation,
15. Uncontrolled massive pleural effusion or massive ascites,
16. Tutelage or guardianship.

Arm A: Specific exclusion criteria for patients with the BRCAness profile in order to receive olaparib

1. Myelodysplastic syndrome/acute myeloid leukemia or with features suggestive of myelodysplastic syndrome (MDS)/ DS)/acute myeloid leukemia (AML),
2. Unable to swallow orally administered medication and gastrointestinal disorders likely to interfere with absorption of the study medication,
3. Any previous treatment with PARP inhibitor, including olaparib,
4. Concomitant use of known strong cytochrome P450, family 3, subfamily A (CYP3A) inhibitors (e.g. itraconazole, telithromycin, clarithromycin, protease inhibitors boosted with ritonavir or cobicistat, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir) or moderate CYP3A inhibitors. The required washout period prior to starting olaparib is 2 weeks,
5. Concomitant use of known strong or moderate CYP3A inducers.
6. Major surgery within 2 weeks of starting study treatment and patients must have recovered from any effects of any major surgery.
7. Previous allogenic bone marrow transplant or double umbilical cord blood transplantation (dUCBT),
8. Whole blood transfusions in the last 120 days prior to entry to the study (packed red blood cells and platelet transfusions are acceptable outside of 28 days prior to study treatment,
9. Known hypersensitivity to the excipients of the olaparib

Arm B/C: Specific criteria for patients without the BRCAness profile and with KRAS mutation in order to receive durvalumab:

1. Prior treatment with any of the following immune checkpoint inhibitor:

   anti-PD-1, anti-PD-L1, anti-PD-L2, or anti-cytotoxic T lymphocyte antigen 4 (CTLA-4) antibody,
2. Active autoimmune disease that has required systemic treatment in the past 2 years; replacement therapy is considered a form of systemic treatment and is not a criterion of exclusion,
3. Any systemic steroid therapy whatever the duration of this corticotherapy,
4. Active or prior documented autoimmune or inflammatory disorders

Arm B/C: Specific exclusion criteria for patients without BRCAness profile and with KRAS-mutated tumors in order to receive selumetinib:

1. Cardiac conditions
2. Documented antecedent history of retinopathy or retinal disorders as known ophthalmologic conditions
3. Patients with any other significant abnormality on ophthalmic examination (performed by an ophthalmologist) should be discussed for potential ineligibility
4. The last palliative radiotherapy seance within 7 days of the first dose of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 307 (Estimated)
Dates: Start 2020-12-07 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
ARM A - Progression free survival (PFS) | at 4 months
  PFS rate at 4 months is defined by the number of patients alive at 4 months from inclusion without PD divided by the total number of patients evaluable at 4 months (dead during 4 months or alive at 4 months with a progressive status available).
ARM B/ C - PFS | Assessed up to 36 months
  PFS is defined as time from randomization into arm B/C to the date of first documented PD RECIST 1.1 and/or iRECIST for arm B and PD RECIST1.1 for arm C or death.

SECONDARY OUTCOMES:
Disease control rate (DCR) | Measured at 16 weeks of maintenance therapy.
  DCR is the percentage of patients who achieve CR, PR, or SD to study treatment (according to RECIST 1.1).
Overall response rate (ORR) | Assessed up to 36 months
  ORR is the number of patients with a best overall response of CR or PR divided by the number of all treated (at least 1 dose of study treatment) patients.
Overall survival (OS) | Assessed up to 36 months
  OS is the time between the date of inclusion into Arm A or Arms B/C and death
Number of participants with treatment-related adverse events | Assessed up to 36 months
  All grade and severe toxicities, according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v5.0
Time to HRQoL score definitive deterioration (TUDD) | At baseline, at every 2 months during treatment, and at the end of treatment visit. Assessed up to 36 months
  TUDD is defined as the time interval between inclusion into Arm A and randomization into Arms B/C and the first occurrence of a decrease in QLQ-C30 score for dimension ⩾5 points compared to baseline HRQoL score without any further improvement in QoL score ⩾5 points or any further available QoL data.

CONTACTS AND LOCATIONS:
Overall Officials: Pascal HAMMEL, MD, Principal Investigator — Hôpital Beaujon
Locations (29):
- France (29):
  - Institut Sainte Catherine, Avignon
  - CHRU Jean Minjoz, Besançon
  - Polyclinique Bordeaux Nord Aquitaine, Bordeaux
  - Centre François Baclesse, Caen
  - Hôpital Beaujon, Clichy
  - GHPSO Site de Creil, Creil
  - Centre Georges François Leclerc, Dijon
  - CHU Dijon, Dijon
  - CHU Grenoble Alpes Hôpital Michallon, Grenoble
  - Hôpital Franco-Britannique, Levallois-Perret
  - CHRU Lille, Lille
  - centre Léon Bérard, Lyon
  - Hôpital Privé Jean Mermoz, Lyon
  - Hôpital Saint Joseph Saint Luc, Lyon
  - CHU La Timone, Marseille
  - Hôpital Européen, Marseille
  - Institut Paoli Calmette, Marseille
  - Hôpital Nord Franche Comté, Montbéliard
  - GH Diaconesses Croix Saint Simon, Paris
  - Hôpital Européen Georges Pompidou, Paris
  - Hôpital Pitié Salpêtrière, Paris
  - Hôpital Saint Antoine, Paris
  - Institut Mutualiste Montsouris, Paris
  - CHU Poitiers, Poitiers
  - CHU Robert Debré, Reims
  - ICO Site de Saint Herblain, Saint-Herblain
  - Centre Paul Strauss, Strasbourg
  - CHU Toulouse IUCT Rangueil, Toulouse
  - Hôpital Trousseau, Tours